CLINICAL TRIAL: NCT00485290
Title: Effect of Meal on Portal and Esophagus Variceal Pressure
Acronym: VIPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No eligible patients were found, the study stopped without including any patients
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Lise Hobolth, MD, Hvidovre Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-KF-2007-0050
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2007-11

CONDITIONS: Cirrhosis; Esophageal Varices
Keywords: cirrhosis, Portal Hypertension, Esophageal Varices, Meal
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices; Hypertension, Portal | interventions — Meals; Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: meal (food intake) — 600 kcal. (16% protein, 49%carbohydrate, 35% fatt)

SUMMARY:
The reason why esophagus varices suddenly rupture and start to bleed is unclear. Food intake increase the hepatic blood flow and the portal pressure, but it is yet unknown if there is also an increase in variceal pressure. The aim of this study is to evaluate the efficacy of a meal on variceal pressure with a non invasive endoscopic measurement device, and compare it with portal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Large Esophageal varices

Exclusion Criteria:

* Treatment with beta-blocking agents
* Respiratory diseases that contradict endoscopy
* Gastric-retention
* Former gastric resection
* Resent sclerotherapy or former banding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
effect of meal on variceal pressure | 30 minutes after the meal

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bendtsen, MD, DMsc., Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark